CLINICAL TRIAL: NCT07214974
Title: Mild Cognitive Impairment Community Screening, Early Detection, and Therapeutic Intervention to Slow Down, or Stop the Progression of the Cognitive Impairment.
Brief Title: Mild Cognitive Impairment Community Screening and Early Intervention Via Stem Cell Therapy and Wearable Brain Computer Interface Device.
Acronym: MCITestCare
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Noah Tech, Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NoahTech; NTMCI0925 (Other: NoahTech, Corp.)
Record Dates: First submitted 2025-09-18; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment (MCI); Early Stages of Cognitive Decline; Alzheimer's Disease Dementia; Alzheimer's Disease Diagnosis; Alzheimer's Disease and Related Dementias; Parkinson's Disease; Parkinson's Disease (PD); Parkinson's Disease With Wearing-off Motor Fluctuations; Dementia (Diagnosis); Dementia MCI (Mild Cognitive Impairment)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Parkinson Disease; Dementia; Disease | interventions — Brain-Computer Interfaces

STUDY DESIGN:
Intervention Model Description: This trial utilizes a parallel assignment model, wherein participants are concurrently randomized to one of four independent intervention arms (control, wellness care, stem cell therapy, or wearable BCI device therapy) for the duration of the study. This design facilitates direct comparisons of efficacy across groups without crossover or sequential elements, ensuring isolation of intervention effects on MCI progression over 5 years.
Who Masked: Participant, Outcomes Assessor
Masking Description: In this double-blind trial, masking is limited to participants and outcomes assessors. No additional parties are masked. Blinding is maintained through the use of identical placebo saline infusions and sham (non-functional) devices across arms, prepared and distributed by an unblinded study coordinator. Intervention delivery is managed by a separate team from the blinded assessors to prevent unblinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Arm 1 (Control) (Placebo Comparator): No active intervention; placebo procedures (e.g., saline infusions or sham devices)
  Interventions: Other: Control - Placebo Comparator
- Arm 2 (Wellness Care) (Active Comparator): Structured wellness programs comprising cognitive training exercises and life
  Interventions: Behavioral: Structured wellness care
- Arm 3 (Stem Cell Therapy) (Experimental): Administration of autologous or allogeneic stem cells via intravenous or
  Interventions: Biological: Stem Cell Therapy - Experimental
- Arm 4 (Wearable BCI Device Therapy) (Experimental): Use of an active non-invasive BCI device for neurofeedback trail
  Interventions: Device: Wearable brain-computer interface devices

INTERVENTIONS:
Behavioral: Structured wellness care — Participants engage in structured wellness programs, including cognitive training exercises (e.g., memory games, problem-solving tasks) and lifestyle counseling focused on diet, physical exercise, sleep hygiene, and stress management. Sham elements may be included for blinding consistency.
  Other Names: Brain-computer Interface (BCI); Stem Cell; wearable BCI
  Arms: Arm 2 (Wellness Care)
Device: Wearable brain-computer interface devices — Participants use an active non-invasive brain-computer interface (BCI) device for neurofeedback training, designed to enhance cognitive function through real-time brain activity monitoring and modulation. Sham (non-functional) devices are provided to other arms for blinding.
  Other Names: stem cell
  Arms: Arm 4 (Wearable BCI Device Therapy)
Biological: Stem Cell Therapy - Experimental — Participants receive administration of autologous or allogeneic stem cells through intravenous or targeted delivery methods aimed at neuroregeneration. Placebo saline infusions are used in other arms to preserve blinding.
  Arms: Arm 3 (Stem Cell Therapy)
Other: Control - Placebo Comparator — Participants receive no active treatment. To maintain blinding, they undergo placebo procedures, such as saline infusions mimicking stem cell therapy or sham (non-functional) devices simulating BCI therapy.
  Arms: Arm 1 (Control)

SUMMARY:
This study aims to evaluate the efficacy of community-based early detection and targeted interventions, including stem cell therapy and wearable non-invasive brain-computer interface (BCI) devices, for Mild Cognitive Impairment (MCI) in adults aged 55 years and older residing in U.S. urban and suburban communities. Primary objectives include assessing improvements in MCI detection rates, cognitive outcomes, and progression delay compared to standard care.

DETAILED DESCRIPTION:
Study Objectives

The primary goal of this investigation is to assess the effectiveness of early MCI detection via community-based screening and subsequent interventions using stem cell therapy and wearable BCI devices. Specific research questions include:

Does community-based screening enhance early detection rates and diagnostic accuracy of MCI relative to conventional clinical practices? Do wellness care interventions post-MCI screening improve cognitive outcomes and delay progression to cognitive decline? What are the epidemiological characteristics and distribution patterns of MCI occurrence in the target population?

Study Design This is a prospective, multicenter, randomized, double-blind, placebo-controlled trial (RCT) designed to minimize bias and ensure methodological rigor.

Eligible participants will be identified through standardized cognitive screening (e.g., Montreal Cognitive Assessment [MoCA]) administered at community facilities and healthcare clinics. Inclusion criteria encompass adults aged ≥55 years with suspected or confirmed MCI, residing in U.S. urban or suburban areas, without contraindications to interventions. Exclusion criteria include severe dementia, active neurological disorders, or inability to provide informed consent.

Participants will be randomized to one of four parallel arms using a computer-generated sequence with stratified block randomization to balance covariates such as age, baseline MCI severity (e.g., MoCA score), and comorbidities. Allocation concealment will be maintained via sequentially numbered, opaque, sealed envelopes managed by an independent data coordinating center.

The intervention arms are defined as follows:

Arm 1 (Control): No active intervention; placebo procedures (e.g., saline infusions or sham devices) will be implemented to preserve blinding where applicable.

Arm 2 (Wellness Care): Structured wellness programs comprising cognitive training exercises and lifestyle counseling (e.g., diet, exercise, and sleep optimization), with sham components for blinding if required.

Arm 3 (Stem Cell Therapy): Administration of autologous or allogeneic stem cells via intravenous or targeted routes, with placebo saline infusions provided to non-stem cell arms.

Arm 4 (Wearable BCI Device Therapy): Use of an active non-invasive BCI device for neurofeedback training, with sham (non-functional) devices distributed to other arms.

Double-blinding will be achieved by ensuring that neither participants nor outcome assessors (e.g., neuropsychologists) are aware of group assignments. Intervention delivery will be handled by a separate team from the assessment personnel to prevent unblinding.

Follow-up evaluations will include periodic cognitive assessments (e.g., MoCA, comprehensive neuropsychological batteries) at baseline, 6 months, 1 year, and annually thereafter for a total duration of 5 years. These will monitor trajectories in cognitive function, MCI progression rates, and secondary endpoints such as quality of life (e.g., via SF-36 questionnaire), neuroimaging biomarkers (e.g., MRI volumetric changes), and biochemical markers (e.g., CSF amyloid-beta levels).

Statistical analysis will adhere to intention-to-treat principles. Inter-group comparisons will employ analysis of variance (ANOVA) or linear mixed-effects models for repeated measures, with adjustments for multiple comparisons (e.g., Bonferroni correction) and covariates. Survival analysis (e.g., Kaplan-Meier curves) will evaluate time-to-event outcomes, such as progression to dementia. Power calculations assume a sample size sufficient to detect a 20% difference in cognitive decline rates with 80% power and α=0.05.

This design facilitates an unbiased assessment of intervention efficacy in mitigating or reversing MCI progression, with potential implications for public health strategies in aging populations.

Last updated: October 03, 2025

ELIGIBILITY:
Inclusion Criteria:

Adults aged 55 years and older Residents of U.S. urban or suburban communities Able to provide informed consent Willing to participate in 3-year follow-up assessments Able to complete cognitive screening assessments Access to transportation for community-based appointments No prior formal diagnosis of dementia

Exclusion Criteria:

Adults under 55 years of age Current diagnosis of moderate to severe dementia Severe psychiatric disorders that would interfere with assessment validity Active substance abuse disorders Severe visual or hearing impairments that cannot be corrected and would prevent assessment completion Terminal illness with life expectancy less than 3 years Current participation in other cognitive intervention research studies Inability to attend follow-up assessments due to geographic relocation plans Significant neurological conditions (stroke, traumatic brain injury, Parkinson's disease) that could confound cognitive assessment Institutionalized individuals (nursing home residents)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-03 (Estimated); Primary Completion 2029-01-03 (Estimated); Study Completion 2030-01-03 (Estimated)

PRIMARY OUTCOMES:
Change in Cognitive Function as Measured by MoCA Score | Baseline, 6 months, 1 year, and annually up to 5 years.
  The primary endpoint is the mean change from baseline in Montreal Cognitive Assessment (MoCA) total score, assessing domains such as memory, attention, language, and executive function. A clinically meaningful improvement is defined as an increase of ≥3 points, while decline indicates progression. This measure evaluates the efficacy of interventions in stabilizing or enhancing cognitive performance.
Rate of Progression to Dementia | Assessed annually over 5 years.
  Proportion of participants progressing from MCI to dementia (e.g., Alzheimer's disease or other forms), diagnosed via DSM-5 criteria and confirmed by neuropsychological evaluation. This assesses intervention effectiveness in delaying or preventing cognitive decline.

SECONDARY OUTCOMES:
Improvement in Neuropsychological Battery Scores | Baseline, 6 months, 1 year, and annually up to 5 years.
  Changes in composite scores from a standardized neuropsychological test battery (e.g., including Rey Auditory Verbal Learning Test for memory, Trail Making Test for executive function, and Boston Naming Test for language). This provides detailed insights into specific cognitive domain improvements.
Change in Quality of Life | Baseline, 6 months, 1 year, and annually up to 5 years.
  Assessed using the Short Form-36 (SF-36) questionnaire, focusing on physical and mental health components. This evaluates the broader impact of interventions on daily functioning and well-being.
Early Detection Rate via Community Screening | Enrollment phase (pre-randomization).
  Proportion of MCI cases identified through community-based MoCA screening compared to historical rates from standard clinical practices in similar populations.

OTHER OUTCOMES:
Epidemiological Characteristics of MCI | Enrollment phase and baseline.
  Descriptive analysis of MCI prevalence, distribution patterns (e.g., by age, sex, urban/suburban residence, comorbidities), and risk factors in the screened cohort. This informs public health strategies.
Safety and Tolerability | Throughout the 5-year study period, reported at each follow-up.
  Incidence and severity of adverse events (e.g., infusion reactions for stem cell therapy, device-related discomfort for BCI), graded per Common Terminology Criteria for Adverse Events (CTCAE).
Adherence to Interventions | Ongoing, summarized annually over 5 years.
  Percentage of completed sessions or device usage compliance, tracked via logs or electronic monitoring, to assess feasibility in real-world settings.

CONTACTS AND LOCATIONS:
Locations (1):
- First Presbyterian Church, Palisades Park, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes